CLINICAL TRIAL: NCT03379337
Title: Pilot Study of a Modular Fluorescent Device With Interchangeable Heads to Identify Oral Diseases
Brief Title: Oral Imaging for Porphyrin Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1603518893
Record Dates: First submitted 2017-12-15; First posted 2017-12-20 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Dental Plaque
Keywords: Imaging
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dental imaging (Experimental): 4 incisors and 4 canine teeth of subjects were imaged with the experimental and the commercial device.
  Interventions: Diagnostic Test: Dental imaging

INTERVENTIONS:
Diagnostic Test: Dental imaging — The target teeth positions for imaging included 4 incisors and all 4 canines. Only the vestibular and interproximal regions were of interest. Images were taken of these target teeth positions regardless of whether or not they exhibited plaque, consisted of full or partial restorations, contained major cracks/fractures, chips, or were missing. Other captured images included any abnormality of the tooth or gum exhibiting red fluorescence physically accessible by the devices.

SUMMARY:
The purpose of this study was to use the principle of fluorescence to identify oral diseases not readily visible to the naked eye. A imaging device with a removable and modular head consisting of arrays of Light Emitting Diodes (LEDs) with differing wavelengths (405nm,450nm or white) was used to image teeth to detect fluorescent biomarkers such as porphyrins associated with poor oral health (plaque). The process utilizes illumination of the teeth and gums using a specific array of LEDs in the visible and near-visible spectrum and is non-invasive. Successful implementation of the device would provide proof-of- concept validation for its use as a safe, rapidly deployable solution to assess oral hygiene.

DETAILED DESCRIPTION:
To use the device, an interchangeable head with a specific LED wavelength was selected (to target a specific oral disease). The optical filter can be exchanged for another if necessary (this is done prior to the subject visit as to not prolong the time of the visit). During operation, LED intensity can be altered using the rotary dimmer switch. The procedure took place during a routine dental visit once consent was obtained. The device was covered in a clear disposable plastic sheath (Consolidated Plastics, Stow, OH) or equivalent sterile disposable camera bag. After both the subject and clinician wore UV protective eyeware, a series of images and videos were taken. These included detailed frames of all 4 incisors and all 4 canines. A video of the camera aperture passing over the select teeth was also taken. Additional images focusing on areas of interest to the clinician were taken, with area of capture and device mode recorded. The total time required to capture all images and video is expected to be approximately 5 minutes. As a control, an Acteon Soprocare a commercial device operating under the same fluorescence principle was also used. Images and video of the aforementioned eight target teeth in each mode were similarly captured for comparison to the test device.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-70. Subjects with identifiable dental diseases must have otherwise healthy tissues/structures in which to control against.

Exclusion Criteria:

Subjects under 18 years of age will not be invited to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
In focus images of all 4 incisors and all 4 canines using devices | 5 minutes for each imaging device used in the study.
  Images of target teeth with imaging devices.

CONTACTS AND LOCATIONS:
Overall Officials: Pratik Shah, Ph.D., Principal Investigator — Massachusetts Institute of Technology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Angelino K, Shah P, Edlund DA, Mohit M, Yauney G. Clinical validation and assessment of a modular fluorescent imaging system and algorithm for rapid detection and quantification of dental plaque. BMC Oral Health. 2017 Dec 28;17(1):162. doi: 10.1186/s12903-017-0472-4. PMID 29284461